CLINICAL TRIAL: NCT03971409
Title: Innovative Combination Immunotherapy for Metastatic Triple Negative Breast Cancer (TNBC): A Multicenter, Multi-Arm Translational Breast Cancer Research Consortium Study
Brief Title: Avelumab With Binimetinib, Sacituzumab Govitecan, or Liposomal Doxorubicin in Treating Stage IV or Unresectable, Recurrent Triple Negative Breast Cancer
Acronym: InCITe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laura Huppert, MD, BA (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Hoosier Cancer Research Network (Other); Array BioPharma (Industry); Pfizer (Industry); Breast Cancer Research Foundation (Other); Johns Hopkins University (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Laura Huppert, MD, BA, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187519; NCI-2019-01531 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TBCRC 047 (Other: Translational Breast Cancer Research Consortium); BRE16-279 (Other: Hoosier Cancer Research Network)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Invasive Breast Carcinoma; Recurrent Breast Carcinoma; Triple-Negative Breast Carcinoma; Unresectable Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — avelumab; binimetinib; utomilumab; liposomal doxorubicin; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- CLOSED TO ENROLLMENT: Arm I (binimetinib, avelumab) (Experimental): Patients will receive a 15-day lead-in of binimetinib, followed by binimetinib PO BID and avelumab IV over 60 minutes every 2 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Binimetinib
- CLOSED TO ENROLLMENT: Arm II (anti-OX40 antibody PF-04518600, avelumab) (Experimental): Patients will receive a 15-day lead-in of anti-OX40 antibody PF-04518600, followed by anti-OX40 antibody PF-04518600 IV over 60 minutes and avelumab IV over 60 minutes every 2 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-OX40 Antibody PF-04518600; Drug: Avelumab
- CLOSED TO ENROLLMENT: Arm III (utomilumab, avelumab) (Experimental): Patients will receive a 15-day lead-in of utomilumab, followed by utomilumab IV over 60 minutes every 4 weeks and avelumab IV over 60 minutes every 2 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Biological: Utomilumab
- Arm A (avelumab, binimetinib, liposomal doxorubicin) (Experimental): Patients receive a 15 day lead-in of binimetinib orally (PO) twice daily (BID) in the absence of disease progression or unacceptable toxicity. Patients then receive binimetinib PO BID on days 1-28, avelumab intravenously (IV) over 60 minutes on days 1 and 15, and liposomal doxorubicin IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Binimetinib; Drug: Liposomal Doxorubicin
- Arm B (avelumab, sacituzumab govitecan) (Experimental): Patients will receive a 15-day lead-in of sacituzumab govitecan given on day -15, followed by sacituzumab govitecan day 8 and day 15 of Cycle (C) 1; day 1,8, and 21 of C2; day 1, 15 and 21 of C3; day 8 and 15 of C4, and schedule continues with two weeks on, one week off for 21-day cycles. Patients also receive 10mg/kg avelumab over 60 minutes on day 1 and day 15 of each 28 day cycle. Cycles repeat in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Sacituzumab Govitecan
- Arm C (avelumab, liposomal doxorubicin) (Experimental): Patients will receive a 15-day lead-in of liposomal doxorubicin, followed by liposomal doxorubicin on Day 1 and 10mg/kg avelumab over 60 minutes on Day 1 and Day 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Liposomal Doxorubicin

INTERVENTIONS:
Biological: Anti-OX40 Antibody PF-04518600 — Given IV
  Other Names: PF-04518600
  Arms: CLOSED TO ENROLLMENT: Arm II (anti-OX40 antibody PF-04518600, avelumab)
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162
  Arms: Arm A (avelumab, binimetinib, liposomal doxorubicin); CLOSED TO ENROLLMENT: Arm I (binimetinib, avelumab)
Biological: Utomilumab — Given IV
  Other Names: PF 05082566; PF 5082566; PF-05082566; PF-2566
  Arms: CLOSED TO ENROLLMENT: Arm III (utomilumab, avelumab)
Drug: Liposomal Doxorubicin — Given IV
  Other Names: Caelyx; Lipodox
  Arms: Arm A (avelumab, binimetinib, liposomal doxorubicin); Arm C (avelumab, liposomal doxorubicin)
Drug: Sacituzumab Govitecan — Given IV
  Other Names: Trodelvy; Sacituzumab Govitecan-hziy
  Arms: Arm B (avelumab, sacituzumab govitecan)

SUMMARY:
This phase II trial studies how well the combination of avelumab with liposomal doxorubicin with or without binimetinib, or the combination of avelumab with sacituzumab govitecan works in treating patients with triple negative breast cancer that is stage IV or is not able to be removed by surgery (unresectable) and has come back (recurrent). Immunotherapy with checkpoint inhibitors like avelumab require activation of the patient's immune system.

This trial includes a two week induction or lead-in of medications that can stimulate the immune system. It is our hope that this induction will improve the response to immunotherapy with avelumab. One treatment, sacituzumab Govitecan, is a monoclonal antibody called sacituzumab linked to a chemotherapy drug called SN-38. Sacituzumab govitecan is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of tumor cells, known as Tumor-associated calcium signal transducer 2 (TROP2) receptors, and delivers SN-38 to kill them. Another treatment, liposomal doxorubicin, is a form of the anticancer drug doxorubicin that is contained in very tiny, fat-like particles. It may have fewer side effects and work better than doxorubicin, and may enhance factors associated with immune response. The third medication is called binimetinib, which may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth, and may help activate the immune system. It is not yet known whether giving avelumab in combination with liposomal doxorubicin with or without binimetinib, or the combination of avelumab with sacituzumab govitecan will work better in treating patients with triple negative breast cancer.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 3 active arms. The three previous study arms are closed to further accrual.

ARM A: Patients receive binimetinib orally (PO) twice daily (BID) for a lead-in period of 15 days in the absence of disease progression or unacceptable toxicity. Patients then receive binimetinib PO BID on days 1-28, avelumab intravenously (IV) over 60 minutes on days 1 and 15, and liposomal doxorubicin IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive sacituzumab govitecan IV on days -15 for a lead-in period in the absence of disease progression or unacceptable toxicity. Patients then receive sacituzumab govitecan day 8 and day 15 of Cycle (C) 1; day 1, 8, and 21 of C2; day 1, 15 and 21 of C3; day 8 and 15 of C4, and the schedule continues with two weeks on, one week off for 21-day cycles which repeat in the absence of disease progression or unacceptable toxicity. Participants also receive avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive liposomal doxorubicin IV over 60 minutes on day -15 for a lead-in period of 15 days in the absence of disease progression or unacceptable toxicity. Patients then receive liposomal doxorubicin IV over 60 minutes on day 15 and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 6 months for a minimum of 1 year. Participants will be followed every 3 months after experiencing disease progression to assess for survival/anti-cancer therapy status until death or 1 year after Cycle 1 Day 1.

PRIMARY OBJECTIVE:

I. Anti-tumor effect of avelumab in combination with different therapeutic agents explored in the sub-protocols of the trial.

SECONDARY OBJECTIVES:

I. Additional anti-tumor effects.

II. Safety and tolerability of avelumab in combination with different therapeutic agents explored in the sub-protocols of the trial.

III. Patient reported outcomes (PRO) between baseline and cycle 3 day 1 across arms.

IV. Longitudinal trends in PRO outcomes across treatment arms.

V. Differences in PRO outcomes for patients who respond compared to those who do not respond.

CORRELATIVE OBJECTIVES:

I. To determine the therapeutic predictive role of the following on clinical outcome as well as changes with induction therapy with either liposomal doxorubicin or targeted agents:

1. PD-L1 expression and immune 'hot-spots'.
2. Tumor infiltrating lymphocyte (TIL)s, and Cluster of differentiation 8 (CD8) and Cluster of differentiation 4 (CD4) positivity in TIL.
3. Human leukocyte antigen (HLA)-A (MHC-I) and HLA-DR (MHC-II), FoxP3, OX40 and OX40L, phosphatase and tensin homologue (PTEN), and MYC expression.
4. Number/levels of expressed predicted class I and class II neoantigens, central memory T-cells and T-cells.
5. Expression of effector/regulatory immune gene, innate PD-1 resistance signature (IPRES), and B cell, T cell, and/or macrophage signatures.
6. Basal or claudin-low molecular subtypes.
7. T cell receptor (TCR) clonality in the tumor and peripheral blood.
8. Genomic mutational burden.

II. To determine if circulating tumor deoxyribonucleic acid (DNA) (ctDNA) results will discriminate pseudo-progression from true progression.

III. To determine if certain genomic alterations detected in tumor tissue or ctDNA are potentially associated with resistance to the tested drug combinations.

IV. To correlate the composition of the pretreatment microbiome with response and secondary endpoints in each arm of the trial.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive binimetinib orally (PO) twice daily (BID) for a lead-in period of 15 days in the absence of disease progression or unacceptable toxicity. Patients then receive binimetinib PO BID on days 1-28, avelumab intravenously (IV) over 60 minutes on days 1 and 15, and liposomal doxorubicin IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive sacituzumab govitecan IV on days -15 and -8 as a lead-in period in the absence of disease progression or unacceptable toxicity. Patients then receive sacituzumab govitecan IV on days 1 and 8 and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive liposomal doxorubicin IV over 60 minutes on day -15. Patients then receive liposomal doxorubicin IV over 60 minutes on day 15 and every 4 weeks thereafter. Patients also receive avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 6 months for a minimum of 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent
2. Subjects >= 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Clinical stage IV invasive breast cancer or unresectable locoregional recurrence of invasive breast cancer meeting the following criteria:

   * Estrogen receptor (ER)/progesterone receptor (PR)-negative (=< 5% cells) by immunohistochemistry (IHC) and human epidermal grow (HER2) negative (by IHC or fluorescence in situ hybridization (FISH))
   * Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria and which can be followed by computed tomography (CT) or magnetic resonance imaging (MRI). A measurable lytic bone lesion(s) and/or skin lesion(s) are allowed. Skin lesions must also be followed by photography with measuring tools within the photograph at each tumor evaluation time point. Ultrasound may be used to follow breast lesions not visible by CT following discussion with Study Chair
   * Amenable to biopsy at the time of study entry
   * Known tumor/immune cell PD-L1 status by any assay
5. Adequate organ function including:

   * Cardiac ejection fraction at or above the institutional lower limit of normal, as assessed by either echocardiogram or multigated acquisition (MUGA) scan
   * Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (may have received growth factor)
   * Platelets >= 100 x 10^9/L
   * Hemoglobin >= 9 g/dL (may have been transfused)
   * Total serum bilirubin =< 1.5 times upper limit of normal (ULN)
   * Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT/serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x ULN (or =< 5 x ULN if liver metastases are present)
   * Serum creatinine =< 1.5 x ULN or estimated creatinine clearance >= 50 mL/min as calculated using the Cockcroft-Gault (CG) equation
   * Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x ULN
   * Amylase =< 1 x ULN testing is only required in patients with a history of pancreatic disorders (Abnormality not of pancreatic origin is allowed)
   * Participants with treated and controlled hypo or hyperthyroidism are eligible.
6. Male and female patients of childbearing potential must agree to use at least two methods of acceptable contraception from 15 days prior to first trial treatment administration until at least 30 days after study participant's final dose of study drug(s)

   * NOTE: Females of childbearing potential are defined as those who are not surgically sterile or post-menopausal (i.e., patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrhoeic for 12 months without an alternative medical cause). Post-menopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone (FSH) level within laboratory reference range for postmenopausal women
7. Patients unable to read/write in English are eligible to participate in the overall study but will not participate in the Patient-Reported Outcome questionnaires throughout the trial.
8. Re-enrollment of a subject that has discontinued the study as a pre-randomization screen failure (i.e., a consented patient who was not randomized and did not receive any study treatment) is permitted. If re-enrolled, the subject must be re-consented. Only the screening procedures performed outside of protocol-specified timing must be repeated; if biopsies and correlative blood samples were already obtained, and patient has not received any systemic anti-cancer therapy since they were obtained, they do not need to be repeated.

Exclusion Criteria:

1. More than 2 lines of chemotherapy in the metastatic setting
2. More than 1 prior line of checkpoint inhibitor therapy in the metastatic setting
3. Prior treatment with sacituzumab, govitecan
4. Concurrent anticancer therapy. Required washout from prior therapies are as follows:

   * Chemotherapy: >= 14 days: antibody drug conjugants administered every 3 weeks require a 3-week washout.
   * Major surgery: >=14 days (provided wound healing is adequate)
   * Radiation: >= 7 days
   * Investigational/biologic therapy (half-life =< 40 hours): >= 14 days
   * Investigational/biologic therapy (half-life > 40 hours): >= 28 days
   * Use of corticosteroids or immunosuppressive medication is exclusionary, except the following in the absence of active autoimmune disease:

     * Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intra-articular, intranasal, and inhaled)
     * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent are permitted
     * Adrenal replacement steroid doses including doses > 10 mg daily prednisone are permitted
     * A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g. CT scan premedication against contrast dye allergy) or for treatment of nonautoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
5. Previous malignant disease other than breast cancer within the last 5 years, with the exception of basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, or low-risk cancers considered curatively treated (i.e. complete remission achieved at least 2 years prior to first dose of study drugs AND additional therapy not required while receiving study treatment)
6. All subjects with central nervous system metastases and/or carcinomatous meningitis, except those meeting the following criteria::

   * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
   * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
   * Subjects must be either off steroids or on a stable or decreasing dose of =< 10 mg daily prednisone (or equivalent)
7. Receipt of any organ transplantation including allogeneic stem-cell transplantation
8. Significant acute or chronic infections including, among others:

   * Known history of testing positive for human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS); testing is not required for this protocol.
   * A history of a positive test for hepatitis B virus (HBV) surface antigen (and/or core antibody) and/or confirmatory hepatitis C virus (HCV) ribonucleic acid (RNA) (if anti-HCV antibody tested positive); testing is not required for this protocol
9. Active autoimmune disease with reasonable possibility of clinically significant deterioration when receiving an immunostimulatory agent, per investigator discretion:

   * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses =< 10 mg or 10 mg equivalent prednisone per day
   * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable
10. History of interstitial lung disease that is symptomatic or which may interfere with the detection or management of suspected drug-related pulmonary toxicity
11. Uncontrolled asthma (defined as having 3 or more of the following features of partially controlled asthma within 28 days prior to starting study treatment: Daytime symptoms more than twice per week, any limitation of activities, any nocturnal symptoms/awaking, need for reliever/rescue inhaler more than twice per week, or known lung function [peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1)] without administration of a bronchodilator that is < 80% predicted or personal best [if known])
12. Current symptomatic congestive heart failure (New York Heart Association > class II), unstable cardiac arrhythmia requiring therapy (e.g. medication or pacemaker), unstable angina (e.g. new, worsening or persistent chest discomfort), uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100mmHg), or known cardiac ejection fraction below the lower limit of institutional normal. Or any of the following occurring within 6 months (180 days) prior to first dose of avelumab: Myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack. (Use of antihypertensive medication to control blood pressure is allowed.)
13. Patients who have neuromuscular disorders that are associated with elevated creatine kinase (CK)
14. History of acute or chronic pancreatitis
15. History or current evidence of retinal vein occlusion (RVO), or current risk factors for RVO including uncontrolled glaucoma, ocular hypertension, history of hyperviscosity, or hypercoagulability syndromes (patients with a history of pulmonary embolism or deep vein thrombosis (DVT) are allowed on study if they are also on anticoagulation as noted in (16) below) ; history of retinal degenerative disease.
16. Requirement of anticoagulant therapy with oral vitamin K antagonists such as Coumadin (warfarin). Low-dose anticoagulants for the maintenance of patency in a central venous access device or the prevention of deep vein thrombosis or pulmonary embolism is allowed. Therapeutic use of low molecular weight heparin or factor Xa inhibitors are allowed provided patients are safely able to interrupt it prior to biopsy procedures.
17. Persisting toxicity related to prior therapy that has not reduced to grade 1 (National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 5.0); however, alopecia and sensory neuropathy grade =< 2 is acceptable
18. Known severe (grade >= 3 NCI-CTCAE v5.0) hypersensitivity reactions to monoclonal antibodies, or history of anaphylaxis
19. Vaccination within 28 days of the first dose of study drugs and while on trial is prohibited, except for administration of inactivated vaccines (for example, inactivated influenza vaccine)
20. Pregnant or breastfeeding females
21. Known current alcohol or drug abuse
22. Prisoners or subjects who are involuntarily incarcerated
23. Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the patient's study physician to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with scheduled visits, treatment schedule, laboratory tests and other study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (BORR) | From treatment initiation until disease progression, an estimated average of 1 year
  BORR is defined as the percentage of patients achieving complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and will be reported for each arm along with 95% two-sided confidence intervals.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From treatment initiation until disease progression, an estimated average of 1 year
  ORR is defined as the percentage of patients achieving complete response (CR) or partial response (PR) assessed by Immune-Related RECIST (iRECIST) and will be reported by arm with 95% two-sided confidence intervals
Clinical Benefit Rate (CBR) | 6 months
  CBR is defined as the percentage of patients achieving complete response (CR), partial response (PR), or stable disease (SD) using RECIST version 1.1 at 6 months and will be reported by arm with 95% two-sided confidence intervals
Median Progression-free Survival (PFS) | From treatment initiation until disease progression, an estimated average of 1 year
  The median duration of progression-free survival in weeks by arm will be estimated using the Kaplan-Meier method with censoring used as needed. Median time to event and corresponding confidence intervals will be reported.
Median Overall Survival (OS) | 12 months
  OS is defined as the time from treatment initiation until disease progression or death, whichever comes first and will be reported by arm with 95% two-sided confidence intervals .
Percentage of participants with treatment-related adverse events | Up to 30 days after completion of study treatment, approximately 13 months
  An unacceptable toxicity is defined as any unexpected and clinically relevant drug-related grade 3 toxicity, or any drug-related grade 4-5 adverse event within the first cycle of therapy assessed via National Cancer Institute CTCAE version 5 criteria. Safety will be evaluated by estimating the percentage of patients who experience a clinically relevant toxicity (both patient and physician reported) for each arm with 95% two-sided confidence intervals.
Change in Quality of Life at 8 Weeks Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Measure | Baseline up to 8 weeks
  Will be measured the PROMIS Global Short Form. Change scores will be compared across treatment arms using one way analysis of variance (ANOVA) with Bonferroni adjustment for post-hoc multiple comparisons. In the instance that distributional assumptions are not valid, Kruskal-Wallis one-way ANOVA will be used with Dunn's adjustment for multiple comparisons.
Change in Quality of Life Over Treatment Duration Assessed by PROMIS Global Health Measure | From baseline until the date disease progression is first observed, an estimated average of 1 year
  Will be measured the PROMIS Global Short Form. Change scores will be compared across treatment arms using one way analysis of variance (ANOVA) with Bonferroni adjustment for post-hoc multiple comparisons. In the instance that distributional assumptions are not valid, Kruskal-Wallis one-way ANOVA will be used with Dunn's adjustment for multiple comparisons.
Change in Symptoms (Self-Reported Toxicities) at 8 Weeks Assessed by Patient-Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Baseline up to 8 weeks
  Will be measured by the PRO-CTCAE criteria . The data will be presented descriptively using summary statistics and graphical representations across time points. Will assess symptom burden using Likert scores. Each attribute will be presented descriptively using summary statistics and graphical representations across time points.
Change in Symptoms (Self-Reported Toxicities) Over Treatment Duration Assessed by PRO-CTCAE | From baseline until the date disease progression is first observed, an estimated average of 1 year
  Will be measured by the PRO-CTCAE criteria . The data will be presented descriptively using summary statistics and graphical representations across time points. Will assess symptom burden using Likert scores. Each attribute will be presented descriptively using summary statistics and graphical representations across time points.
Change in Ability to Participate in Social Roles and Activities at 8 Weeks Assessed by PROMIS | Baseline up to 8 weeks
  The data will be presented descriptively using summary statistics and graphical representations across time points. Change scores will be compared across treatment arms using one way ANOVA with Bonferroni adjustment for post-hoc multiple comparisons. In the instance that distributional assumptions are not valid, Kruskal-Wallis one-way ANOVA will be used with Dunn?s adjustment for multiple comparisons.
Change in Ability to Participate in Social Roles and Activities Over Treatment Duration Assessed by PROMIS | From baseline until the date disease progression is first observed, an estimated average of 1 year
  The data will be presented descriptively using summary statistics and graphical representations across time points. Change scores will be compared across treatment arms using one way ANOVA with Bonferroni adjustment for post-hoc multiple comparisons. In the instance that distributional assumptions are not valid, Kruskal-Wallis one-way ANOVA will be used with Dunn?s adjustment for multiple comparisons.
Change in Treatment Satisfaction at 8 Weeks Assessed by the Treatment Satisfaction Questionnaire for Medication (TSQM) | Baseline up to 8 weeks
  Will be assessed by TSQM Questionnaire. Change scores will be compared across treatment arms using one way ANOVA with Bonferroni adjustment for post-hoc multiple comparisons. In the instance that distributional assumptions are not valid, Kruskal-Wallis one-way ANOVA will be used with Dunn?s adjustment for multiple comparisons.
Change in Treatment Satisfaction Over Treatment Duration Assessed by the TSQM | From baseline until the date disease progression is first observed, an estimated average of 1 year
  Will be assessed by TSQM Questionnaire. Change scores will be compared across treatment arms using one way ANOVA with Bonferroni adjustment for post-hoc multiple comparisons. In the instance that distributional assumptions are not valid, Kruskal-Wallis one-way ANOVA will be used with Dunn?s adjustment for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Huppert, MD, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (12):
  - O'Neal Comprehensive Cancer Center, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago Medicine Comprehensive Cancer Center, Evergreen Park, Illinois
  - Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No